CLINICAL TRIAL: NCT03916445
Title: Resilience and Quality of Life in Patients With Gynaecological Carcinomas and Chronic Gynaecological Diseases: A Pilot Study
Brief Title: Resilience and Quality of Life in Patients With Gynaecological Carcinomas and Chronic Gynaecological Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00366
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Gynecologic Disease; Gynecologic Cancer
MeSH Terms: conditions — Genital Diseases, Female | interventions — Connor-Davidson Resilience Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gynecological cancer: all patients having a consultation doctor during the recruiting time
  Interventions: Other: Connor Davidson Resilience Scale (CD-RISC 10)
- chronic gynecological disease: all patients having a consultation doctor during the recruiting time
  Interventions: Other: Connor Davidson Resilience Scale (CD-RISC 10)

INTERVENTIONS:
Other: Connor Davidson Resilience Scale (CD-RISC 10) — questionnaires about resilience (Connor Davidson Resilience Scale(CD-RISC 10)) and quality of life (EQ-5D-5L)
  Other Names: EQ-5D-5L

SUMMARY:
The intended pilot project aims at evaluating the feasibility and acceptability of questionnaires about resilience and quality of life in two different patient groups (either with a gynaecological carcinoma ora chronic gynaecological disease). The results provided by this pilot study will build the basis of an upcoming, larger project including these questionnaires and the main objective of assessing resilience. More precisely, the study aims at answering the following questions. How is the overall resilience and quality of life in the target population at one assessment point? Are the instruments used in this pilot feasible for the target population when assessing resilience and quality of life?

ELIGIBILITY:
Inclusion Criteria:

* female,
* >18 years old,
* german speaking

exclusion criteria:

- insufficient study language skills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with a chronic gynecological disease or a gynaecological carcinoma, currently treated at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
resilience measured by questionnaire | up to 1 year
  Total Score of the resilience questions is 0 to 40, 10 subscales from 0 to 4 (summed up for total score), the higher the score the better the resilience

SECONDARY OUTCOMES:
quality of life measured by questionnaire | up to 1 year
  Questions about Quality of life: Total score 0-25, 5 subscales 0 to 5 (summed up for total score), the higher the score the lower is Quality of life.

OTHER OUTCOMES:
quality of life measured by VAS in the questionnaire | up to 1 year
  visual analogue scale (VAS) about Feeling healthy: Score 0 to 100 the higher the score the better is Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Viola Heinzelmann-Schwarz, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitätsspital Frauenklinik, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No